CLINICAL TRIAL: NCT02201719
Title: Norwegian Adenomyosis Study: Pathophysiology, Peristalsis, Expression Profiling and Diagnostics, Part I
Brief Title: Norwegian Adenomyosis Study I
Acronym: NAPPED I
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Tina Tellum, Medical Doctor, Oslo University Hospital
Other Study IDs: 2014/637a
Record Dates: First submitted 2014-07-02; First posted 2014-07-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Dysmenorrhea; Chronic pelvic pain; Infertility; Sensitivity histology; womens health; junction zone
MeSH Terms: conditions — Adenomyosis; Dysmenorrhea; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hysterectomy Adenomyosis: Adenomyosis present
- Hysterectomy no adenomyosis: Adenomyosis not present

SUMMARY:
Adenomyosis is characterized by the appearance of endometrial cells in the muscular layer of the uterus. It affects about 15-20% of the female population.

The symptoms of adenomyosis are heavy menstrual bleedings and painful menstruation (dysmenorrhea) and in addition chronic pelvic pain. Subfertility and infertility have been correlated with adenomyosis.

Parity, age and uterine abrasion increase the risk of adenomyosis. Hormonal factors such as local hyperestrogenism and elevated levels of prolactin have been identified, but autoimmune and mechanical factors are also hypothesized.

Regarding treatment, the most effective measure is hysterectomy. As this is a very drastic measure in younger women, levonogestrel-releasing intrauterine devices, Gonadotropin releasing hormone (GnRH)-analogues, Danazol, uterine embolization and endometrial ablation have been tried, but studies are few in number, retrospective, and have small sample sizes.

Adenomyosis has so far not been subject to extensive research efforts. The pathogenesis of adenomyosis remains still unclear, there are not many satisfying treatment options and diagnostics include mostly magnetic resonance imaging (MRI) and histology.

The investigators designed a series of 3 studies with a broad approach in understanding adenomyosis. This is part 1.

NAPPED-1: comparison of 3D-transvaginal ultrasound with MRI and histology in the diagnostic of adenomyosis

DETAILED DESCRIPTION:
Diagnosis of Adenomyosis with 3D and 2D transvaginal ultrasound. Prospective study of a consecutive series of 101 patients that are scheduled for hysterectomy and suffer from bleeding disorders, chronic pelvic pain, dysmenorrhea or dyspareunia. All patients will undergo transvaginal 2D- ultrasound, 3D-ultrasound and power doppler (PD)-ultrasound (TVU), magnetic resonance imaging of the pelvic organs (MRI) and hysterectomy.

We will investigate the specificity and sensitivity of 3D and 2D transvaginal ultrasound in the diagnosis of adenomyosis and compare data with MRI and histopathology, which is the gold standard by today. In addition, we will collect anamnestic information that might point to risk factors or connections to prior obstetrical complications and medicine use. In our study the pathologist will not be blinded to our ultrasound findings, and we want to investigate if this will raise the sensitivity of histology findings of adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 30 - 50 years old
* scheduled for vaginal, abdominal or laparoscopic total hysterectomy
* one or more of the following clinical symptoms: bleeding disorders (menorrhagia, irregular bleeding, hypermenorrhoea), chronic pelvic pain, dysmenorrhoea, or dyspareunia
* junction zone definable

Exclusion Criteria:

* postmenopausal women,
* pregnancy
* gynecological cancer
* GnRH analog therapy or systemic hormone therapy in the last three months prior to hysterectomy
* junctional zone not identifiable

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women referred to our clinic and volunteering to participate and that are registrated in Norway with a norwegian social security number.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference in sensitivity and specificity of 3D TVU and MRI; in percentage points (%) | within 4 weeks after 3D TVU
  Sensitivity and specificity of 3D TVU in the diagnosis of adenomyosis compared to MRI.

SECONDARY OUTCOMES:
Positive and negative predictive value of 3D TVU in percent (%) | within 17 weeks after 3D TVU
  Positive and negative predictive value of 3D TVU in diagnosis of adenomyosis. The histological examination is the end-point because it is still regarded to be the gold-standard in diagnosis of adenomyosis.
Difference in sensitivity and specificity of 3D TVU and 2D TVU; in percentage points (%) | within 17 weeks after 3D TVU
  The sensitivity and specificity of 3D TVU in the diagnosis of adenomyosis will also be compared to 2D TVU, in addition to MRI (see primary outcome measure).
Difference in max. thickness of junction zone, in millimeters (mm) | post ovulatory in any menstruational cycle prior to surgery, within 4 weeks after 3D TVU
  Compares measurements of junction zone made by 3D TVU and MRI.
Prevalence of sub- and infertility, percent (%) | at time of enrollment
  Questionnaire-based investigation. Prevalence of sub- and infertility in their medical history of the study population.
Difference in sensitivity and specificity of 3D TVU and histopathology; in percentage points (%) | within 17 weeks after 3D TVU
  The sensitivity and specificity of 3D TVU in the diagnosis of adenomyosis will also be compared to 2D TVU, in addition to MRI (see primary outcome measure) and histopathology, which is still the gold standard.
Prevalence of miscarriages, in percent (%) | at time of enrollment
  Questionnaire-based investigation. Prevalence of miscarriages in the medical history of the study population.
Prevalence of previous gynecological surgeries, in percent (%) | at time of enrollment
  Questionnaire-based investigation. Prevalence of previous gynecological surgical interventions in the medical history of the study population.
Prevalence of previous obstetrical complications, in percent (%) | menarche to time of enrollment
  Questionnaire-based investigation. Prevalence of previous obstetrical complications in the medical history of the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Marit Lieng, PhD, MD, Principal Investigator — Oslo University Hospital, Ullevål
Locations (1):
- Department of Gynecology, Oslo University Hospital Ullevål, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Tellum T, Nygaard S, Skovholt EK, Qvigstad E, Lieng M. Development of a clinical prediction model for diagnosing adenomyosis. Fertil Steril. 2018 Oct;110(5):957-964.e3. doi: 10.1016/j.fertnstert.2018.06.009. PMID 30316443